CLINICAL TRIAL: NCT03761446
Title: The Role of Type 2 Diabetes on Skeletal Muscle Atrophy and Recovery Following Bed Rest in Older Adults
Acronym: REST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TRIMD 1330040
Record Dates: First submitted 2018-10-30; First posted 2018-12-03 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Muscle Atrophy; Aging; Sedentary Behavior; Pre-diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Muscular Atrophy; Sedentary Behavior; Glucose Intolerance | interventions — Bed Rest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Older adults with pre-diabetes or type 2 Diabetes (Experimental): Male and female older adults between the ages 60-80 with pre-diabetes or type 2 diabetes
  Interventions: Behavioral: Bed rest
- Older adults without pre-diabetes or Type 2 Diabetes (Experimental): Male and female older adults between the ages 60-80 without pre-diabetes or type 2 diabetes
  Interventions: Behavioral: Bed rest

INTERVENTIONS:
Behavioral: Bed rest — The participant will remain in bed rest for 10 complete days.

SUMMARY:
The goal of this study is to determine the impact of pre-diabetes and type 2 diabetes on muscle atrophy during a period of bed rest and recovery of muscle mass, strength, and physical function following bed rest.

DETAILED DESCRIPTION:
Older adults with type 2 diabetes experience an accelerated rate of sarcopenia, which is the deterioration in muscle mass, strength and physical performance. Periods of disuse caused by illness or hospitalization cause rapid loss of muscle mass and strength, which negatively impact physical function upon re-ambulation. The impact of type 2 diabetes on acute muscle atrophy and recovery from disuse is a critical issue that has not been investigated.

The overall objectives of this study are to employ highly innovative methods in muscle biopsy specimens in order to decipher the temporal sequence by which mitochondrial dysfunction and lipotoxicity in older adults with pre-diabetes and type 2 diabetes impact atrophy and recovery of muscle mass, strength and physical function following bed rest. Older adults with and without pre-diabetes/type 2 diabetes will complete 10 days of strict bed rest followed by 4 weeks of ambulatory recovery. During bed rest muscle biopsies will be collected to determine mitochondrial function and lipid profile. During the recovery period the recovery of muscle mass, strength and physical function will be determined.

ELIGIBILITY:
Inclusion Criteria

1. Participant must be male or female between the ages of 60 and 80 years of age.
2. Participant has pre-diabetes or type 2 diabetes and is only taking DPP-4 inhibitors, Sulfonylureas and/or Metformin therapy (but not Insulin, injectable incretin mimeticsSGL2 inhibitors, and Thiazolidinedione's), and has an A1C < 8.0.

   1. Pre-Diabetics are defined as having an HgbA1c of greater than or equal to 5.7% and less 6.5%, or a fasting glucose of greater than or equal to 100 mg/dl and less than 126 mg/dl or has a glucose of greater than or equal to 140 mg/dl and less than 200mg/dl at the 2 hour blood draw during OGTT
   2. The non-diabetic control group is defined as having an HgbA1c of less than 5.7%, a fasting glucose of less than 100 mg/dl and a glucose level less than 140 mg/dl at the 2hr blood draw during the OGTT.
3. Participant must have renal function with an estimated glomerular filtration rate (eGFR) > 45 ml/min/1.73m2 determined at screening.
4. Participant's triglyceride level is < 350 mg/dl and LDL cholesterol is ≤ 150 mg/dl at screening.
5. Participants must be non-smokers. Non-smokers as defined by not smoking any tobacco or using nicotine-containing products and not using vape pens or vaporizers within 3 months prior to screening.
6. Participant states willingness to follow protocol as described, including consumption of study product per protocol, the prescribed activity level and completing any forms needed throughout the study.
7. Participant has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board/Independent Ethics Committee, and provided Health Insurance Portability and Accountability Act authorization (HIPAA) or other privacy authorization prior to any participation in study.

Exclusion Criteria

1. Participant has type 1 Diabetes.
2. BMI > 40.0 kg/m2
3. Participant is actively pursuing weight loss and/or lifestyle changes.
4. Participant has a history of pressure ulcers.
5. Participant has a stated history of Deep Vein Thrombosis (DVT), pulmonary embolism, or a known hypercoagulable condition, or other clotting or bleeding disorders.
6. History of gastrointestinal or intracranial hemorrhage.
7. History of stroke or cerebrovascular accident.
8. Recent history of major trauma (within 3 months).
9. Thrombocytopenia (of any cause) or hyperkalemia (K > 5.0) on screening laboratory assay. May repeat lab value per PI discretion.
10. Untreated or poorly controlled hypertension (SBP > 150, DBP > 95), or hypotension (SBP <100 DBP <60)
11. Participant has a TSH greater than or equal to 10mIU/L.
12. Participant has current infection (requiring prescription antimicrobial or antiviral medication, or hospitalization), or corticosteroid treatment (with the exception of inhaled or topical steroids) in the last 3 months prior to screening visit.
13. Participant is currently taking anti-inflammatory medication or has anti-inflammatory medication in the 1 weeks prior to screening (including over the counter formulations; e.g. Aleve, Motrin, ibuprofen, naproxen).
14. Participant has had surgery requiring > 2 days of hospitalization in the last 1 month prior to screening visit.
15. Participant has an active malignancy or autoimmune disease.
16. Participant has current significantly impaired liver function in the opinion of the study PI (mild asymptomatic fatty liver is acceptable), or hepatic enzyme tests are ≥ 2.5 times normal limit.
17. Participant has a chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV.
18. Participant is an amputee and/or has presence of partial or full artificial limb.
19. Participant has had a significant cardiovascular event (e.g. myocardial infarction, stroke) ≤ 6 months prior to screening visit; or stated history of congestive heart failure; or participant has evidence of cardiovascular disease assessed during the ECG at screening. In the event of a positive stress test, participants are referred to their primary care physician. If the electrocardiogram (ECG) is determined to be a false positive, participant may be allowed to participate in study after confirmatory records obtained.
20. Participant has a history of, or currently has uncontrolled severe diarrhea, nausea or vomiting.
21. Participant has an obstruction of the gastrointestinal tract, inflammatory bowel disease, short bowel syndrome or other forms of gastrointestinal disease such as stage III or above gastroesophageal reflux disease, gastroparesis, peptic ulcer disease, celiac disease, intestinal dysmotility, diverticulitis, ischemic colitis and bariatric surgery.
22. Participant cannot abstain from alcohol for the pre bed rest and bed rest portion of the study. For the recovery portion of the study the participant must agree to consume no more than 1 glass of wine (4-5 oz) or bottle of beer (12 oz) /day.
23. Participant cannot refrain from taking medications/dietary supplements/herbals or substances that could modulate glucose metabolism (other than oral hypoglycemic medications), or are considered anabolic, or reduce weight (fat mass), or that may interact with low-molecular weight heparin or induce hypo- or hyper-coagulable state, in the opinion of the PI or medical provider, starting one week prior to enrollment and over the entire course of the study. These include progestational agents (except prescribed birth control), steroids, growth hormone, dronabinol, marijuana, calcium-beta-hydroxy-betamethylbutyrate (CaHMB), free amino acid supplements and dietary supplements to aid weight loss.
24. Participant has a mini-Mental State Examination score < 21.
25. Subjects who fulfill any of the contraindications for MRI; examples include metal implants, devices, paramagnetic objects contained within the body and excessive or metal-containing tattoos.
26. Unable to participate in MR or DEXA assessments due to physical limitations of equipment tolerances (e.g., MRI bore size and DEXA 450-pound weight limit) claustrophobia, or based on Investigator's judgment at screening.
27. Participant has a sensitivity or allergy to lidocaine.
28. Participant has a sensitivity or allergy to heparin, enoxaparin, or other low molecular weight heparin.
29. History of allergy to pork products or any component of the formulation of low-molecular weight heparin for dosing.
30. History of heparin induced thrombocytopenia.
31. Hemoglobin < 10.0 g/dL for females; < 11.0 g/dL for males; or participant has clinically significant signs/symptoms of anemia in the opinion of the PI or medical provider.
32. Concomitant medications with known contraindication or interaction with low-molecular weight heparin (including anti-platelet agents, anti-coagulant agents, non-steroidal anti-inflammatory drugs)
33. Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete the study.
34. Participant experiences symptoms of claudication. Symptoms include cramping pain in the legs and/or difficulty walking.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Leg Lean Mass | Pre and Post Bed Rest and following 4 weeks of ambulatory recovery
  Determined by DXA (dual energy x-ray absorptiometry)
Mitochondrial Respiration | Pre and Post Bed Rest
  Determined by high resolution respirometry in permeabilized muscle fiber bundles

SECONDARY OUTCOMES:
Insulin Sensitivity | Pre and Post Bed Rest
  Determined by hyperinsulinemic euglycemic glucose clamp
Physical function | Pre and Post Bed Rest
  Determined by short physical performance battery

CONTACTS AND LOCATIONS:
Overall Officials: Paul Coen, PhD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No